CLINICAL TRIAL: NCT04147507
Title: Effect of Relaxing Music on Blood Pressure and Resting Heart Rate Among Pre-hypertensive Young Adults
Brief Title: Effect of Relaxing Music on Blood Pressure and Resting Heart Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Imtiyaz Ali Mir, Principal Investigator, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMFB1012
Record Dates: First submitted 2019-10-29; First posted 2019-11-01 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Prehypertension; Blood Pressure; Resting Heart Rate
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental)
  Interventions: Other: Passive Music Therapy
- Control (Other): Life style Modification.
  Interventions: Behavioral: Control

INTERVENTIONS:
Other: Passive Music Therapy — Music group (N=15) will receive listen to music therapy passively for 20 minutes/day, 5 days/week for 4 weeks, along with lifestyle modifications. Music therapy will be provided via headphones in an isolated quiet non-disrupted room, with room temperature maintained between 20-22 degree Celsius and having medium light intensity. Participants would be instructed to listen to music with eyes closed in sitting position, back supported in comfortable position on a chair. The participants will be given 5 minutes' rest in sitting position before and after each music therapy session.
  Arms: Music Therapy
Behavioral: Control — Control group (N=15) would receive only lifestyle modification. Handout of lifestyle modification according to the Seventh Joint National Committee (JNC VII) report guidelines will be given to all participants. Participants would be instructed to not participate in any form of physical activity and to focus only on two components from the guideline which includes practice the DASH eating plan (diet rich in fruits and vegetables, low fat dairy or unsaturated fat) and limit the daily sodium intake (less than 100 mmol per day).
  Arms: Control

SUMMARY:
Prehypertention is defined as systolic blood pressure between 120 and 139 mmHg and/or diastolic blood pressure between 80 and 89 mmHg. People with prehypertension have the higher risk to develop hypertension compared to people with normal blood pressure (normotensive) especially when getting old, therefore prehypertension is known for preliminary stage of hypertension. Framingham Heart Study have shown the progression rate from prehypertension to hypertension was as high as 19% over 4 years. Prehypertension will also lead to abnormality of the cardiovascular system. Thus it is very important to identify the prehypertension at early stage, so that steps can be taken to slow down the progression to hypertension and to normalize the blood pressure level. Minimal reduction in blood pressure produce a large benefit to human health, as stated in JNC (Joint National Committee) VII report, a 5mmHg decrease in systolic blood pressure would be able to reduce as much as 9% mortality rate caused by coronary heart disease, 14% mortality related to stroke, and 7% decrease in all-cause mortality. Previous studies have focused on effect of music therapy in hypertensive elderly, prehypertensive pregnant women, prehypertensive elderly but no research has been conducted on prehypertensive young adults. In addition, prehypertension increase risk of developing cardiovascular disease, thus early intervention is needed to prevent the progression of prehypertension to hypertension status and normalize the blood pressure level.

DETAILED DESCRIPTION:
Quota sampling will be used as the sampling method. Investigators would recruit 30 participants for this study.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure between 120 to 139 mmHg
* Diastolic blood pressure between 80 to 89 mmHg
* Not having any hearing impairment and able to listen to music using headphone
* Willing to participate in this study

Exclusion Criteria:

* Under influence of any medication that would affect the concentration
* Systolic Blood pressure of less than 120 or more than 140 mmHg
* Diastolic blood pressure of less than 80 or more than 90 mmHg

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants with prehypertension.
Enrollment: 30 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure change is being measured | At baseline (before intervention) and post intervention (end of 4 weeks)
Diastolic Blood Pressure change is being measured | At baseline (before intervention) and post intervention (end of 4 weeks)
Resting Heart Rate change is being measured | At baseline (before intervention) and post intervention (end of 4 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers